CLINICAL TRIAL: NCT00833313
Title: Gene Expression Profiling in Subjects With Postoperative Atrial Fibrillation After Cardiac Surgery (GENEXPRO Surg)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Jochen Daniel Muehlschlegel, MD, Associate Professor, Brigham and Women's Hospital
Other Study IDs: 2008-P000896
Record Dates: First submitted 2009-01-05; First posted 2009-02-02 (Estimated); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Atrial Fibrillation
Keywords: Atrial fibrillation; Gene expression; Genetic
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Atrial tissue sample
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Atrial biopsy — Biopsy of left atrial free wall and possibly left atrial appendage

SUMMARY:
Atrial fibrillation is a type of irregular heartbeat that is common after having heart surgery. There may be many different reasons why some people get atrial fibrillation after their heart surgery. These reasons may include that a person is older or that he/she is taking certain types of medications before surgery. Genes may also be a reason. Genes contain the material passed from parent to child that determines the make-up of the body and mind. For example, some genes control the color of your hair or eyes. Some people may have genes that make it more likely for them to get atrial fibrillation after their heart surgery. This research project is being done to find out if the cells of people who develop atrial fibrillation after heart surgery are different from the cells in people who do not develop atrial fibrillation after surgery.

DETAILED DESCRIPTION:
Atrial fibrillation is a type of irregular heartbeat that is common after having heart surgery. There may be many different reasons why some people get atrial fibrillation after their heart surgery. These reasons may include that a person is older or that he/she is taking certain types of medications before surgery. Genes may also be a reason. Genes contain the material passed from parent to child that determines the make-up of the body and mind. For example, some genes control the color of your hair or eyes. Some people may have genes that make it more likely for them to get atrial fibrillation after their heart surgery. This research project is being done to find out if the cells of people who develop atrial fibrillation after heart surgery are different from the cells in people who do not develop atrial fibrillation after surgery.

This study seeks to identify regulatory events in atrial myocyte transcription and translation that are altered by germline variation

ELIGIBILITY:
Inclusion Criteria:

* Age 20-99 years
* Undergoing cardiac surgery

Exclusion Criteria:

* Prior cardiac surgery
* chest radiation
* recent chemotherapy

Ages: 20 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients undergoing cardiac surgery
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2008-08 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Gene expression | Immediate

CONTACTS AND LOCATIONS:
Overall Officials: Jochen D Muehlschlegel, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Result] Sigurdsson MI, Saddic L, Heydarpour M, Chang TW, Shekar P, Aranki S, Couper GS, Shernan SK, Muehlschlegel JD, Body SC. Post-operative atrial fibrillation examined using whole-genome RNA sequencing in human left atrial tissue. BMC Med Genomics. 2017 May 2;10(1):25. doi: 10.1186/s12920-017-0270-5. PMID 28464817
- [Result] Sigurdsson MI, Saddic L, Heydarpour M, Chang TW, Shekar P, Aranki S, Couper GS, Shernan SK, Seidman JG, Body SC, Muehlschlegel JD. Allele-specific expression in the human heart and its application to postoperative atrial fibrillation and myocardial ischemia. Genome Med. 2016 Dec 6;8(1):127. doi: 10.1186/s13073-016-0381-1. PMID 27923400